CLINICAL TRIAL: NCT00569985
Title: A Pilot Study of Safety and Feasibility of Stem Cell Therapy for Aids Lymphoma Using Stem Cells Treated With a Lentivirus Vector-Encoding Multiple Anti-HIV RNAs
Brief Title: Gene Therapy-Treated Stem Cells in Treating Patients Undergoing Stem Cell Transplant for Intermediate-Grade or High-Grade AIDS-Related Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04047; CHNMC-04047; NCI-2012-00437 (Registry Identifier: NCI CTRP); 04047 (Other: City of Hope Medical Center)
Record Dates: First submitted 2007-12-07; First posted 2007-12-10 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Lymphoma
Keywords: AIDS-related diffuse large cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; HIV-associated Hodgkin lymphoma; Treatment Experienced
MeSH Terms: conditions — Lymphoma | interventions — Carmustine; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (autologous HCT) (Experimental): CONDITIONING: Patients receive carmustine IV over 1-2 hours on days -7 to -5, etoposide IV over 4 hours on day -4, and cyclophosphamide IV on day -2. TRANSPLANTATION: Patients undergo autologous hematopoietic stem cell transplantation comprising lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells and non-bound CD34+ cells IV on day 0.
  Interventions: Biological: lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells; Drug: carmustine; Drug: cyclophosphamide; Drug: etoposide; Procedure: autologous hematopoietic stem cell transplantation

INTERVENTIONS:
Biological: lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells — Undergo autologous hematopoietic stem cell transplantation comprising lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells and non-bound CD34+ cells
  Other Names: lentivirus-transduced hematopoietic progenitor cells
Drug: carmustine — Given IV
  Other Names: BCNU; BiCNU; bis-chloronitrosourea
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Procedure: autologous hematopoietic stem cell transplantation — Undergo autologous hematopoietic stem cell transplantation comprising lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells and non-bound CD34+ cells

SUMMARY:
This pilot clinical trial studies biological therapy in treating patients with acquired immune deficiency syndrome (AIDS)-related lymphoma undergoing stem cell transplant. Giving chemotherapy before a stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. After treatment, stem cells are collected from the patient's blood and stored. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. Giving biological therapy as part of the stem cell transplant may be more effective in treating patients with AIDS-related lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and feasibility of using lentivirus-transduced hematopoietic progenitor cells (HPCs) (lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells) in the setting of autologous hematopoietic cell transplantation (HCT) for treatment of AIDS related lymphoma. The safety of the of the genetically modified product used in the transplant procedure will be assessed by monitoring each subject for adverse events (procedure related toxicity); absolute neutrophil count (ANC)/platelet engraftment (sustained recovery); and evidence of replication competent vector or vector recombination with the human immunodeficiency virus (HIV) quasi-species present in the patient.

II. To determine the quantity and duration of vector-marked peripheral blood cells and to characterize: the duration and level of gene marking and expression of the anti-HIV ribonucleic acids (RNAs) in these transduced cells, and the characterization of the integration sites of vector sequences in circulating cells if there is a clinical syndrome suggestive of a clonal expansion of hematopoietic cells. In addition, the feasibility of the process will be assessed based on the results of the release testing of the transduced cells prior to injection into the patient.

III. To determine whether the design of the vector prevents vector mobilization and rescue by wild-type HIV-1. IV. To measure the effect of HIV infection on the presence of HIV-resistant blood cells as measured by genetic marking for vector sequences before and after antiviral treatment interruption.

OUTLINE:

CONDITIONING: Patients receive carmustine intravenously (IV) over 1-2 hours on days -7 to -5, etoposide IV over 4 hours on day -4, and cyclophosphamide IV on day -2.

TRANSPLANTATION: Patients undergo autologous hematopoietic stem cell transplantation comprising lentivirus vector rHIV7-shI-TAR-CCR5RZ-transduced hematopoietic progenitor cells and non-bound cluster of differentiation (CD)34+ cells IV on day 0. After completion of study treatment, patients are followed up every 2 weeks for 3 months; at 4, 6, 8, 10, 12, 18, and 24 months; every 6 months for 3 years; and then annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive at or before the time of lymphoma diagnosis
* Anti-HIV chemotherapy; subjects must be on a multi-drug regimen (excluding azidothymidine) and have an HIV viral load < 50,000 copies/ml by reverse transcriptase-polymerase chain reaction (RT-PCR) at the time of study enrollment
* Subjects must agree to have their anti-HIV regimen temporarily stopped, and then all subjects will stop antiretroviral therapy (ART) for approximately 7 days at the time they start filgrastim (G-CSF) post-chemotherapy for peripheral blood progenitor cell (PBPC) mobilization and until the mobilization is complete; in addition, if/when the CD4 counts return to a level of 450/mm^3 with undetectable HIV levels in blood, the subjects will undergo an analytic treatment interruption for an indefinite period not to exceed 6 months
* Karnofsky performance status >= 70%
* Biopsy proven intermediate grade or high-grade non-Hodgkin's lymphoma, including plasmablastic lymphoma, primary effusion lymphoma, or biopsy-proven Hodgkin's lymphoma (entities as defined in the World Health Organization [WHO] classification); tissue histology will be reviewed at the City of Hope; patients with prior marrow involvement must demonstrate =< 10% involvement pre-stem cell collection
* No psychosocial conditions that would hinder study compliance and follow-up
* Pretreatment serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic pyruvic transaminase (SGPT) =< 2.5 x institutional upper limit of normal (ULN)
* Serum bilirubin =< 2.5 x institutional ULN
* Patients who are hepatitis C virus (HCV) antibody positive or hepatitis B virus (HBV) surface antigen positive must be free of clinical evidence of cirrhosis that would otherwise make them ineligible for HCT, as determined by the Principal Investigator (PI) in consultation with the Gastrointestinal Service at City of Hope; patients with HBV and ongoing evidence of viral replication may require therapy prior to receiving high-dose chemotherapy
* Serum creatinine =< 2 x institutional ULN and a 24 hour urine creatinine clearance >= 60 cc/min
* Prothrombin time (PT)/partial thromboplastin time (PTT) =< 2 x normal
* Forced expiratory volume in 1 second (FEV1) or diffusion capacity of the lung for carbon monoxide (DLCO) >= 50% predicted
* Left ventricular ejection fraction (LVEF) >= 50% (by 2-dimensional [2-D] echocardiogram or multigated acquisition scan [MUGA]); absence of cardiomyopathy, congestive heart failure or dysrhythmia
* If the subject is female and of child-bearing potential, subject must have negative serum or urine pregnancy test within 7 days of treatment with research agent; men with partners of child-bearing potential and women of child-bearing potential, must be willing to use medically effective birth control methods, e.g. contraceptive pill, condom, or diaphragm and continue this for one year post HCT
* Subjects must be on a prophylactic regimen for Pneumocystis carinii pneumonia, or agree to begin such treatment, if the CD4 counts are =< 200

ELIGIBILITY CRITERIA (HODGKIN LYMPHOMA) - First or greater relapse after initial complete remission; or partial remission; or induction failure that responds to salvage therapy with stable disease, partial remission, or complete remission (i.e. chemosensitive disease)

ELIGIBILITY CRITERIA (NON-HODGKIN LYMPHOMA):

- First complete remission with high risk features as specified by the International Prognostic Index, or Relapse after prior complete remission; partial remission; or induction failure that responds to salvage therapy with stable disease, partial remission, or complete remission (i.e. chemosensitive disease)

SECONDARY ELIGIBILITY CRITERIA:

* Subjects must complete both the therapeutic and research phases of the G-CSF mobilization of peripheral blood progenitor cells and
* Subjects must have collected at least 5 x 10^6 CD34+ cells/kg for the research phase of the collections

Exclusion Criteria:

* Presence of detectible HIV-1 that has C-X-C chemokine receptor type 4 (CXCR4)-tropism
* Any symptomatic bacteria or fungal infection
* AIDS related opportunistic infections within the past year for which treatment has been unsuccessful would be considered exclusionary but on a case-by-case basis as determined by the PI
* Active cytomegalovirus (CMV) retinitis or other active CMV-related organ dysfunction; patients with a history of treated CMV infection are not excluded
* Relapse of Pneumocystis carinii pneumonia within the past year
* Intractable and severe diarrhea, defined as > 1500 cc diarrheal fluid per day, or diarrhea causing persistent severe electrolyte abnormalities or hypoalbuminemia
* Other AIDS-related syndromes, infectious or otherwise, if perceived to cause excessive risk for morbidity post-HCT, as determined by the PI
* History of grade III hemorrhagic cystitis due to prior cyclophosphamide chemotherapy
* Pregnant or nursing women
* Any prior malignancy, except those treated with curative intent that are five years from treatment or cervical and anal squamous cell cancers or superficial basal cell and squamous cell cancers of skin
* Active central nervous system (CNS) lymphoma; patients with a history of positive cerebrospinal fluid cytology that has become negative with intrathecal chemotherapy are eligible
* Abnormal cytogenetics not related to the lymphoma
* History of myocardial infarction or congestive heart failure
* Any history of HIV-associated encephalopathy; dementia of any kind; seizures in the past 12 months; any perceived inability to directly provide informed consent (note: consent may not be obtained by means of a legal guardian)
* Any medical or physical contraindication or other inability to undergo HPC-apheresis (HPC-A) collection
* Elevated amylase or lipase SGOT, SGPT > 2.5 x the institutional ULN
* Serum bilirubin > 2.5 x ULN
* Any other laboratory value for complete blood count (CBC) and chemistry panel > 2 x ULN

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2007-06; Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Safety of treatment using the National Cancer Institute (NCI) hematologic Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 15 years post stem cell infusion
  The toxicities observed after each stem cell infusion will be summarized in terms of type (organ affected or laboratory determination such as ANC), severity (by NCI CTCAE version 3 and nadir or maximum values for the laboratory measures), time of onset (i.e., course number), duration, and reversibility of outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.
Survival of shI-TAR-CCR5RZ-marked cells in the peripheral blood, demonstrated by presence of transgene by Q-PCR using primers specific for rHIV7-shI-TAR-CCR5RZ in serial samples of peripheral blood | 24 months post stem cell infusion
Determination of RNA transgene expression in samples of peripheral blood mononuclear cells (PBMCs) or marrow before and after infusion, analyzed by Northern blotting/hybridization | Day 1 post stem cell infusion
  For detection of the shRNA, we will use a quantitative real-time PCR assay.
Analysis of vector rescue by HIV | 15 years post stem cell infusion
  Integration analysis will be performed only if there is a clinical syndrome that suggests clonal expansion of hematopoietic cells. In that situation, the method of insertion site location will use a linear amplification mediated (LAM)-PCR technique. If positive vector sequences are found in the plasma, confirmation of vector rescue will be done by isolation of HIV and subsequent HIV sequencing.
Ability to obtain suitable numbers of lentiviral vector treated HPC-A | Day 2 post apheresis
  The number and type of cells will be determined by fluorescence-activated cell sorting (FACS) analysis of the final cell product. Target number for untransduced cells in the final therapeutic cell product is 2.5 x 10^6 CD34+ cells/kg. Minimum target number of CD34+ cells for transduction is 5 x 10^6/kg and in the final transduced cell product, the number of CD34+ cells must be >= 2.0 x 10^6 CD34+ cells/kg with total viability >= 70%. The relative or absolute number of transduced CD34+ cells will be determined.
Determination of replication competent lentivirus (RCL) and HIV-1/vector recombination | 15 years post stem cell infusion

CONTACTS AND LOCATIONS:
Overall Officials: Amrita Y. Krishnan, MD, Study Chair — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States